CLINICAL TRIAL: NCT06407596
Title: High-intensity Laser Therapy (HILT) or Conventional Combined Physical Therapy in the Management of Hemiplegic Shoulder Pain ; Randomized Controlled Trial
Brief Title: HILT or Conventional Combined Physical Therapy, in the Management of Hemiplegic Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: is E2-22-1902
Record Dates: First submitted 2024-03-29; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Hemiplegic Shoulder Pain; Hemiplegia; Physical Therapy; High Intensity Laser
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1: high intensive laser (Experimental): HILT was applied 3 times per week, totaling 9 sessions for three weeks.
  Interventions: Device: high intensity laser
- group 2: TENS+Ultrasound (Experimental): tens+us used combined. 5 times per week. total 15 sessions for three weeks
  Interventions: Device: tens+us

INTERVENTIONS:
Device: high intensity laser — 3 times per week, for 9 sessions
  Arms: group 1: high intensive laser
Device: tens+us — 5 times per week, total 15 sessions for 3 weeks
  Arms: group 2: TENS+Ultrasound

SUMMARY:
Background: Hemiplegic shoulder pain is one of the most common complications after a stroke. There are many treatment strategies for this complication. High-intensity laser therapy (HILT) is a new treatment option, and we aimed to compare the effectiveness of conventional electrotherapy agents and HILT in this study.

Patients and methods: Participants (N = 42) were randomized into the HILT (n = 21) and TENS+US (n = 21) groups. Group 1 received 3 sessions of HILT per week for 3 weeks in addition to a therapeutic exercise program that performed 5 sessions per week for 3 weeks. Group 2 received conventional physical therapy and a therapeutic exercise program for HSP of 5 sessions per week for 3 weeks. Patients were assessed before and after treatment on the on the 6th week for radiological evaluation with ultrasonography and for clinical parameters with VAS, AMAT, MRS, and FIQ scores.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed case of HSP,
* Age ≥18,
* First-ever unilateral stroke,
* Visual analog scale (VAS) ≥30 mm,
* Time since stroke ≥6 months,
* Time since last local intervention treatment >6 months.

Exclusion Criteria:

* A history of shoulder pain prior to stroke;
* An unstable medical condition or uncontrolled systemic diseases (such as respiratory failure, congestive heart failure, liver and kidney dysfunction, or any other disorders affecting neuromuscular function);
* Bilateral hemiplegia;
* Cardiac pacemakers;
* Disturbance of awareness, severe visual and cognitive impairment, Mini-Mental State Examination score: <23 points

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
visual analog scale | before treatment(baseline), after treatment
  pain level, between 0-10, 0 is no pain, 10 is very severe pain
arm motor ability test | before treatment(baseline), after treatment
  this scale asses the upper extremity motor function improvement and daily living activity level , between 0 is the worst score, mean is cant do/use, 5 is the best score.(between 0-5)
functional indepandance measures | before treatment(baseline), after treatment
  functional capacity assessment scale;and despite indepandance of daily living activity 0-126, high score is better function
modified ranking scale | before treatment(baseline), after treatment
  determines the patient's addiction level and evaluates disability; the score is between 0 and 6, where 0 is complete well-being, 5 is very severe disorder and 6 is full dependency

SECONDARY OUTCOMES:
ultrasonographic imaging | before treatment(baseline), after treatment
  muscle-skeletal ultrasonographic imaging;ultrasonographic findings; SA-SD bursitis, Bicipital tenosynovitis, Tendinosis, Cortical irregularity, Partial rupture, Total rupture, ACJ joint hypertrophy, Calcific tendinitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No